CLINICAL TRIAL: NCT00911898
Title: A Phase 1 and Pharmacologic Study of MM-111 in Patients With Advanced, Refractory Her2 Amplified, Heregulin Positive Cancers
Brief Title: A Study of MM-111 in Patients With Advanced, Refractory Her2 Amplified, Heregulin Positive Cancers
Acronym: Monotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-111-01-100
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Her2 Amplified Solid Tumors; Metastatic Breast Cancer
Keywords: Her2 amplified solid tumors; Breast Cancer; Her3/ErbB3; Bispecific Antibody
MeSH Terms: conditions — Breast Neoplasms | interventions — MM-111

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MM-111 (Experimental)
  Interventions: Drug: MM-111

INTERVENTIONS:
Drug: MM-111 — For Phase 1: Dose-escalation cohorts, drug is administered weekly via IV

SUMMARY:
This study is an open-label Phase 1 trial of MM-111.

DETAILED DESCRIPTION:
Phase 1: Patients with any solid tumor type may be enrolled to evaluate the safety and tolerability of MM-111.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced cancer that is:

  * HER2 amplified (IHC 2+ or greater) based on archived tumor evaluation
  * Heregulin positive based on a study required fresh biopsy sample performed at screening and confirmed by central laboratory
* Patients must have blocks of archived formalin-fixed, paraffin-embedded tumor tissue available for sectioning and immunohistochemical staining
* Patient's cancer must have recurred or progressed following standard therapy, have not responded to standard therapy, or for which no standard therapy exists.
* Patients must be >= 18 years of age
* Patients or their legal representatives must be able to understand and sign an informed consent
* Patients may have measurable or non-measurable tumor(s)
* Patients should have ECOG Performance Score (PS) 0 or 1
* Patients must have adequate bone marrow reserves as evidenced by:

  * Absolute neutrophil count (ANC) >= 1,500/uL and
  * Platelet count >= 100,000/uL
  * Hemoglobin >= 9 g/dL
* Patients must have tumor tissue amenable to biopsy
* Patients must be willing to undergo biopsy prior to treatment to MM-111

Exclusion Criteria:

* Patients for whom potentially curative antineoplastic therapy is available
* Patients who are pregnant or lactating
* Patients with an active infection or with an unexplained fever greater than 38.5 C during screening visits or on the first scheduled day of dosing. (At the discretion of the investigator, patients with tumor fever may be enrolled)
* Patients with untreated and/or symptomatic primary or metastatic CNS malignancies (patients with CNS metastases who have undergone surgery or radiotherapy, whose disease is stable, and who have been on a stable dose of corticosteroids for at least 2 weeks prior to the first scheduled day of dosing will be eligible for the trial
* Patients with known hypersensitivity to any of the components of MM-111 or who have had hypersensitivity reactions to fully human monoclonal antibodies (patients with a history of hypersensitivity to trastuzumab, a humanized antibody, are not excluded)
* Patients with known HIV, hepatitis B or C (if patients have previously been treated for C and have undetectable viral loads, they can be considered eligible for the trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muralidhar Beeram, MD, Principal Investigator — The START Center for Cancer Care
Locations (4):
- United States (4):
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Indiana University (IUPUI), Indianapolis, Indiana
  - Fox Chase Center, Philadelphia, Pennsylvania
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MM-111
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MM-111
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 61.0 [30 to 82]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Secondary Outcome: To Determine the Clinical Activity of MM-111 in Patients Based on Objective Response Rate (ORR), Duration of Response (DoR), Progression Free Survival (PFS), and 16 & 24-week Clinical Benefit Rate (CBR)
Time Frame: December 2011
Reporting Status: Not Posted

2. Secondary Outcome: To Explore the Role Functional Imagining (FDG-PET CT Scan), as a Predictor of Clinical Activity
Time Frame: December 2011
Reporting Status: Not Posted

3. Primary Outcome: Maximum Tolerated Dose (MTD) or Maximum Feasible Dose
Description: The Maximum Tolerated Dose (MTD) was defined as the highest dose level in which a DLT is experienced by fewer than two patients in a cohort of 3 - 6 patients. If a DLT is observed in at least two patients in a cohort of 3 - 6 patients, the MTD will be determined to have been exceeded and an additional three patients (up to a total of six) are to be treated at the next lower dose level.
Time Frame: 28 days
Measure: Number; unit: mg/kg
Groups:
- MM-111: All participants
Arm/Group | MM-111
Number analyzed (Participants) | 20
mg/kg | NA [4.4 to 8.0] — MTD was not attained as no patients experienced a dose limiting toxicity.

ADVERSE EVENTS:
Arm/Group | MM-111
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MM-111 (N=20)
Disease Progression (General disorders) | 1
Peural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Acute viral myocarditis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MM-111 (N=20)
Fatigue (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No